CLINICAL TRIAL: NCT02071771
Title: DAILIES® AquaComfort Plus® Toric - Comparative Assessment of Visual and Mechanical Performance
Brief Title: Visual Assessment of DAILIES® AquaComfort Plus® for Astigmatism as Compared to 1-DAY ACUVUE® MOIST® for Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M-14-007
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Astigmatism
Keywords: DACP Toric; DAILIES® AquaComfort Plus®; Astigmatism; Toric
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DACP T, Then 1DAM A (Other): Nelfilcon A toric contact lenses worn first, with etafilcon A toric contact lenses worn second. Each product worn bilaterally on a daily wear, daily disposable basis for 10 days.
  Interventions: Device: Nelfilcon A toric contact lenses; Device: Etafilcon A toric contact lenses
- 1DAM A, Then DACP T (Other): Etafilcon A toric contact lenses worn first, with nelfilcon A toric contact lenses worn second. Each product worn bilaterally on a daily wear, daily disposable basis for 10 days.
  Interventions: Device: Nelfilcon A toric contact lenses; Device: Etafilcon A toric contact lenses

INTERVENTIONS:
Device: Nelfilcon A toric contact lenses
  Other Names: DACP Toric; DAILIES® AQUACOMFORT PLUS® TORIC
Device: Etafilcon A toric contact lenses
  Other Names: 1-DAY ACUVUE® MOIST® for Astigmatism

SUMMARY:
The purpose of this study is to evaluate functional vision associated with rotational stability at blink of DAILIES® AquaComfort Plus® Toric (DACP T) compared to 1-DAY ACUVUE® MOIST® for Astigmatism (1DAM A).

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent document;
* Wear toric soft contact lenses within the protocol-specified range;
* Cylinder equal or higher than -0.75 diopters (D) in both eyes;
* Have an acceptable fit with both study contact lenses;
* Willing to wear lenses for a minimum of 5 days per week, 6 hours per day, every day, if possible;
* Best corrected visual acuity (BCVA) of 20/30 Snellen;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any ocular infection, inflammation, abnormality, or disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications that would contraindicate contact lens wear, as determined by the investigator;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Require presbyopic correction;
* Any ocular condition observed during examination at the enrollment visit;
* History of herpetic keratitis, ocular surgery or irregular cornea;
* Pregnant or lactating;
* Participation in any clinical trial within 30 days of the enrollment visit;
* Currently wearing Focus® DAILIES® Toric or 1-DAY ACUVUE® MOIST® for Astigmatism;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, EMEA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the US and 1 study center located in the UK.
Pre-assignment Details: This reporting group includes all enrolled participants, as treated. Note: 2 participants randomized to DACP T were exited prior to dispense due to unacceptable fit (1) and unavailable lens power (1).
Period: Period 1: First 10 Days
Arm/Group | DACP T, Then 1DAM A | 1DAM A, Then DACP T
Started | 41 | 39
Dispensed | 39 | 39
Completed | 39 | 39
Not Completed | 2 | 0
Not completed — Unacceptable lens fit | 1 | 0
Not completed — Unavailable lens power | 1 | 0
Period: Period 2: Second 10 Days
Arm/Group | DACP T, Then 1DAM A | 1DAM A, Then DACP T
Started | 39 | 38 (One participant completed Period 1 but did not start Period 2 due to unacceptable fit with DACP T.)
Completed | 39 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis group includes all randomized subjects who had no major protocol violations excluding those who met the critical deviation criteria as specified in the Deviations and Evaluability Plan.
Groups:
- Overall: Nelfilcon A and Etafilcon A toric contact lenses worn during Period 1 and Period 2, as randomized, in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: High Contrast Time Controlled Visual Acuity (TCVA) at Day 10
Description: TCVA test was performed at 4 meters under high illumination (90%) using a Landolt ring test. For each acuity level, a series of single rings with gaps in one of four directions was presented and the percentage of correctly identified rings constituted the score. TCVA was measured in VA units and a higher TCVA value indicates an improvement in visual acuity. Both eyes contributed to the analysis.
Time Frame: Day 10, each product
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: VA units
Groups:
- DACP T: Nelfilcon A toric contact lenses worn bilaterally during Period 1 or Period 2 on a daily wear, daily disposable basis for 10 days.
- 1DAM A: Etafilcon A toric contact lenses worn bilaterally during Period 1 or Period 2 on a daily wear, daily disposable basis for 10 days.
Arm/Group | DACP T | 1DAM A
Number analyzed (Participants) | 69 | 69
VA units | 0.02 (0.94) | 0.04 (0.92)

2. Secondary Outcome: Lens Oscillation at Blink at Day 10
Description: Lens oscillation (rotational stability of the lens on the eye) at blink was video-recorded. Digital images were used to measure the rotational characteristics of the lenses and objectively measure the amplitude of the lens oscillation. A higher value indicates greater lens movement on the eye. This outcome measure was collected at one site only.
Time Frame: Day 10, each product
Population: This analysis group includes all randomized subjects at the UK site with data at visit who had no major protocol violations excluding those who met the critical deviation criteria as specified in the Deviations and Evaluability Plan.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | DACP T | 1DAM A
Number analyzed (Participants) | 38 | 38
degrees
  Right Eye | 2.1 (1.0) | 2.7 (1.1)
  Left Eye | 2.1 (1.0) | 2.5 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (5 months). This analysis group includes all subjects exposed to investigational product based on treatment-specific exposure, as reported by the subject or observed by the investigator.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects whether or not related to the medical device. Note: 2 subjects were exposed to DACP T but not dispensed.
Groups:
- DACP T: Nelfilcon A toric contact lenses worn bilaterally on a daily wear, daily disposable basis for 10 days.
- 1DAM A: Etafilcon A toric contact lenses worn bilaterally on a daily wear, daily disposable basis for 10 days.
Arm/Group | DACP T | 1DAM A
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/78
Other Adverse Events (participants affected / at risk) | 0/79 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.